CLINICAL TRIAL: NCT01304576
Title: Orientation Agnosia: Neuropsychological Evaluation, Associated Symptoms, Clinical and Anatomical Correlations
Brief Title: Orientation Agnosia: Clinical and Anatomical Study
Acronym: AGNORIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2009/126/HP; number ID RCB 2009-A01005-52 (Other: Afssaps)
Record Dates: First submitted 2010-08-23; First posted 2011-02-25 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Cerebrovascular Disorders; Brain Lesions
Keywords: stroke; parietal lesions
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient with right parietal lesions (Experimental)
  Interventions: Behavioral: Neuropsychological testing; Other: MRI
- patient with left parietal lesions (Active Comparator)
  Interventions: Behavioral: Neuropsychological testing; Other: MRI

INTERVENTIONS:
Behavioral: Neuropsychological testing — Experimental test about orientation agnosia and standard neuropsychological tests.
Other: MRI — Cerebral MRI

SUMMARY:
The area of the brain responsible of visuospatial processing data and more specifically the orientation of an object or image is located in parietal lobe, especially on the right side. A dysfunction of this region would result in a disorder of recognition of the orientation of objects and images that the investigators call orientation agnosia. Several isolated cases are reported in the literature but to the investigators knowledge deficit has never been systematically searched, or put into perspective compared to other neuropsychological deficits. Moreover, the precise location of the lesion responsible for such a disorder remains uncertain. The objectives of this study are (1) detect the existence of orientation agnosia in case of right parietal lesion, and (2) to improve the understanding of such a deficit allowing better management of this disorder.

DETAILED DESCRIPTION:
Idem

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* french language
* right parietal lesion on cerebral imaging (CT-scan is sufficient), including stroke,arterial malformation, isolated tumoral lesion
* informed consent

Exclusion Criteria:

* previous neurological history except non complicated migraine and stabilized epilepsia without seizure since 5 years
* previous psychiatric history except depression without hospitalization > one week or anxiety with maximum one anxiolytic treatment
* drug or alcohol abuse
* severe cranial traumatism
* other severe chronic pathology
* psychotropic medication other than a hypnotic or an anxiolytic at low doses without dose modification for at least one month
* visual impairment
* motor or sensory deficit sufficient to render impossible neuropsychological tests
* patient without judicial or administrative liberty
* measure of legal protection or no capable to express their consent
* pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
orientation agnosia evaluation | 1 week to 6 months (average)
  orientation agnosia test

SECONDARY OUTCOMES:
associated clinical symptoms especially apraxia | 1 week to 6 months (average)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MARTINAUD, Doctor, Principal Investigator — Service de neurologie et centre mémoire de ressources et recherche
Locations (1):
- CHU de Rouen - Hôpitaux de Rouen, Rouen, Haute-Normandie, France

REFERENCES:
- [Derived] Carlier J, Le Goff F, Pouliquen D, Bliaux E, Bioux S, Gerardin E, Cruypeninck Y, Segobin S, Savoure A, Martinaud O. Evaluation of the cognitive outcome after out-of-hospital cardiac arrest: The role of thalamus. Eur J Neurosci. 2023 Jun;57(11):1892-1912. doi: 10.1111/ejn.15978. Epub 2023 May 8. PMID 37066486